CLINICAL TRIAL: NCT06430749
Title: Clinical Trial of Evaluating Efficacy and Safety for Percutaneously Prostate Cancer Lesion Targeted Microwave Tissue Coagulation as Prostate Functional Preservation
Brief Title: Targeted Microwave Tissue Coagulation for Prostate Cancer
Acronym: MicroPro2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Osamu Ukimura (Other)
Responsible Party: Sponsor-Investigator, Osamu Ukimura, Professor, Kyoto Prefectural University of Medicine
Organization: Kyoto Prefectural University of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTREC-S220202; jRCTs052240015 (Other: Japan Registry of Clincal Trials)
Record Dates: First submitted 2024-05-21; First posted 2024-05-28 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave Tissue Coagulation Arm (Experimental): The Minimally invasive microwave coagulation surgery will be performed under general anesthesia for aiming to be provided total 65 patients.
  Interventions: Device: Microtaze

INTERVENTIONS:
Device: Microtaze — Targeted Microwave Tissue Coagulation
  Other Names: AFM-712

SUMMARY:
This clinical trial is to provide a minimally invasive treatment option in which the targeted prostate cancer tissue is killed by microwave only in the specific area of cancer "that should be treated for saving of life," while leaving a portion of the normal prostate tissue that is not cancerous. This treatment is named "focal therapy" for "clinically localized prostate cancer." As this new treatment aims to treat only the specific prostatic area of cancer, it is different from the invasive conventional treatment to remove the entire prostate gland. The goal is both to control the known cancer by treating only the cancerous area and to maintain the quality of life (QOL) by leaving the other normal prostate tissue and its surrounding organs intact, resulting in the prevention of urinary leakage and sexual dysfunction as complications.

DETAILED DESCRIPTION:
This trial will provide ultrasound-guided targeted microwave tissue coagulation of known cancer lesions in patients diagnosed with clinically localized prostate cancer, and it will assess efficacy and safety endpoints for up to six months post-operatively. This trial will also assess patient quality of life (QOL).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who have a single lesion of PI-RADS category 3 or 4 lesion on MRI image at enrollment and which is proved as a Gleason score 7 or 8 on histopathology of the prostate needle biopsy at enrollment; or, patients who have a single lesion of PI-RADS category 4 or 5 lesion on MRI image at enrollment and which is proved as a Gleason score 6 or 7 on histopathology of the prostate needle biopsy at enrollment
2. Patients with prostate cancer that is clinical stage T2c or lower (T1a-T2cN0M0) according to the TNM Classification as determined during enrollment
3. Patients between the ages of 20 and 85 when providing consent to participate in this trial
4. Patients from whom consent is obtained prior to enrollment in this trial

Exclusion Criteria:

1. Patients to have a lesion identified as PI-RADS category 4 or 5 on MRI images at enrollment and which is a diameter of less than 10 mm and Gleason score of 6 on the histopathology of the prostate needle biopsy at enrollment (the lesion is referred to as 'non-target lesions') (the diameter of the lesion is defined as the longer one of the lesion diameter identified on MRI images at enrollment or the tumor length as measured on histopathology of prostate needle biopsy)
2. Patients to have 4 or more non-target lesions (non-target lesions are defined as the lesions defined in exclusion criterion 1, or lesions with PI-RADS category 3 on MRI image at enrollment and Gleason score 6 on biopsy at enrollment)
3. Patients to have a lesion with PI-RADS category 5 on MRI image at enrollment and Gleason score 8 on histopathology of prostate needle biopsy at enrollment (the lesion is referred 'excluded lesions')
4. Patients with a serum prostate-specific antigen (PSA) level over 20 ng/ml during enrollment
5. Patients in whom the distance from the target prostate cancer lesion to the rectum is 10 mm or less on MRI images (coronal or sagittal) obtained during enrollment
6. Patients who have received an antiandrogen for benign prostatic hyperplasia prior to enrollment
7. Patients who have received an antiandrogen for benign prostatic hyperplasia prior to enrollment
8. Patients who have undergone surgery, drug therapy, or radiation therapy for prostate cancer prior to enrollment
9. Patients with active multiple cancers
10. Patient who wear a pacemaker
11. Patients for whom MRI scans are contraindicated
12. Patients in whom transrectal ultrasound cannot be performed for some reason, such as a constricted rectum
13. Patients with a prothrombin time<50% or platelet count<60,000/mm3 during enrollment
14. Patients deemed to be ineligible by an investigator

Ages: 20 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants achieving disappearance of cancer | 6 months
  Disappearance of cancer is defined with the following criteria:
  1. A 50% or greater reduction from the preoperative serum PSA level.
  2. A reduction of PI-RADS category of the targeted prostate cancer lesion down to 3 or lower (including 'difficult to judge' and 'change after treatment') on MRI images.
  3. No cancer tissue in histopathological examination from the targeted prostate cancer lesion via a needle biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Osamu Ukimura, Professor, Principal Investigator — Kyoto Prefectural University of Medicine
Locations (1):
- Kyoto Prefectural University of Medicine, Kyoto, Japan

IPD SHARING:
Plan to Share IPD: No